CLINICAL TRIAL: NCT07006116
Title: Caregiver Bootcamp: Mastering the First Hundred Days
Brief Title: Caregiver Bootcamp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Carolyn Clevenger, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007427; 2P30AG064200-06 (NIH)
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Dementia
Keywords: Caregiver; Dementia; Person living with dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The investigators will enroll caregivers in six cohorts of 8 each to participate in this Stage Ib clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Synchronous/asynchronous online course Participants (Experimental): The program will combine 5 weekly small group (8 participants) 90-120-minute online sessions with asynchronous instructional materials delivered 2-4 days in between sessions.
  A time suited to all for the synchronous sessions will be identified. The research team will provide instructions for accessing the weekly sessions and asynchronous segments, and mail out supplemental course materials. The team will track online attendance, and the Canvas platform will enable them to monitor each individual's viewing of the asynchronous materials.
  Interventions: Other: Synchronous/asynchronous online course

INTERVENTIONS:
Other: Synchronous/asynchronous online course — * Synchronous weekly 90-120-minute-long sessions that will be conducted on a videoconferencing platform (i.e., Zoom). If participants miss a synchronous session.
  * Asynchronous online course: available segments of the online course with asynchronous instructional materials delivered 2-4 days in between sessions, and supplemental course materials that will be received by mail.

SUMMARY:
This study will assess the preliminary efficacy of a synchronous/asynchronous psychoeducation program designed to promote caregiving mastery in the immediate time period after a dementia diagnosis. It will also study the effects on caregiver and care recipient well-being.

DETAILED DESCRIPTION:
The Caregiver Bootcamp program will employ psychoeducational methods (expert instruction, expectation of active learning by participants, debriefing and coaching linked to participant reports of application of strategies and principles) to enhance the proposed mechanism of action of the intervention, the enhancement of caregiving mastery - the individual's self-acknowledgement of self-efficacy for coping with the stresses of the new caregiving role.

The program is meant to provide basic orientation to the situation: recognize the reality of the condition; understand the shifts in mindset that the immediate situation demands; begin to recognize the shift in responsibility that will have to occur; and take practical steps to prepare for the future. The program will combine 5 weekly small group 90-120-minute online sessions with asynchronous instructional materials delivered 2-4 days in between sessions.

ELIGIBILITY:
Inclusion Criteria:

1. over the age of 21;
2. care partner/caregiver for a family or friend who has received a diagnosis of a form dementia from a healthcare provider in the last 6 months;
3. has access to an electronic device and/or access to broadband internet; and
4. able to speak and understand English. Caregivers are not required to be co-located with the care recipient.

Exclusion Criteria:

* considering moving the PLWD to an institutional setting within the next 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver sense of mastery | Baseline, 1 and 3-months post-intervention
  The seven-item personal mastery scale developed by Pearlin and Schooler is used to measure mastery. All items are rated on a four-point scale: 1 = strongly agree; 2 = agree; 3 = disagree; to 4 = strongly disagree. Total scores ranged from 7 to 28, with higher scores indicating higher levels of mastery.
Change in caregiver self-efficacy: symptom management scale | Baseline, 1 and 3-months post-intervention
  This outcome will be assessed with Likert scale questions. Includes 6 questions, each scored on a 0-10 scale. Total possible score range is 0-60, with higher score correlating with better study outcome.
Change in caregiver self-efficacy: support services scale | Baseline, 1 and 3-months post-intervention
  This outcome will be assessed with Likert scale questions. Includes 4 questions, each scored on a 0-10 scale. Total possible score range is 0-40, with higher score correlating with better study outcome.
Change in caregiver self-efficacy: medication management scale | Baseline, 1 and 3-months post-intervention
  This outcome will be assessed with Likert scale questions. Includes 5 questions, each scored on a 0-10 scale. Total possible score range is 0-50, with higher score correlating with better study outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Clevenger, RN, DNP, Principal Investigator — Emory University
Locations (1):
- Nell Hodgson Woodruff School of Nursing, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with controlled access for general research use as allowed by participants' informed consent and contingent on a requesting institution's Institutional Review Board approval and investigators' approved data sharing plan
Time Frame: Scientific data will be made available no later than the on-line publication of the main findings from investigators' final dataset and all other generated scientific data will be shared no later than the end of the project award. Study data for the trial will be stored in the Emory Roybal Center repository for at least 5 years.
Access Criteria: De-identified data from Roybal-supported trials will be available to qualified researchers through a data sharing agreement that will be fully consistent with NIH data sharing policies and applicable laws and regulations as well as official policies and practices established by the Emory Roybal Center.